CLINICAL TRIAL: NCT02876497
Title: Study of Trans-tissular Migration of Macrophages Associated to Human Breast Cancer
Acronym: Macrophages
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 16 SEIN 03
Record Dates: First submitted 2016-07-28; First posted 2016-08-23 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study arm (Experimental)
  Interventions: Other: Define macrophages migration mode

INTERVENTIONS:
Other: Define macrophages migration mode — Archival tumor samples analysis and blood sample testing

SUMMARY:
Surgical samples of human primitive breast: Representative and various surgical samples of human primitive breast carcinoma in terms of histological type. Moreover, healthy tissue from the same patient will be analysed in parallel. Adjacent normal epithelial structures will be defined as at least 5 mm away from the tumor and histologically normal in appearance.

Isolation, differentiation of human monocyte-derived Macrophages (Mphs) and determination of the Macrophage (Mph) migration mode : Human Mphs will be differentiated from blood monocytes isolated from the same patient than the tumor sample. Blood samples will be obtained following standard ethical procedures.

DETAILED DESCRIPTION:
Surgical samples of human primitive breast: In order to use human samples from the anatomo-pathological laboratory collection, several statements will be signed and coordinated by the legal department of Centre National de Recherche Scientifique (CNRS) and Institut National de la Santé et de la Recherche Médicale (INSERM) in accordance with Centre Hospitalier Universitaire (CHU). Representative and various surgical samples of human primitive breast carcinoma in terms of histological type (no special type, lobular etc …), grade, tumor size (except tumor less than 1 cm for having enough material), hormone receptor status, HER2 status and index of proliferation will be prospectively analysed. Moreover, healthy tissue from the same patient will be analysed in parallel. Adjacent normal epithelial structures will be defined as at least 5 mm away from the tumor and histologically normal in appearance, as independently determined by a clinical pathologist.

All clinical characteristics of the patients will be collected : age at diagnosis, body mass index, nulliparous status or not, pre-peri- or post- menopausal status, systemic adjuvant treatment in terms of hemotherapy, tailored therapy and local treatments. Moreover all histo-pathological characteristics of the infiltrative primary breast carcinoma will be determined by team 2 :histological type (no special type, lobular etc …), grade Scarff-Bloom et Richardson (SBR), tumor size, hormone receptor status (estrogen and progesterone receptor), HER2 status (overexpression/amplication), index of proliferation (count of mitosis and antigen KI67), presence or not of embole vascular, presence or not of in-situ carcinoma and nodal status. For the human breast tissue cohort, the amounts of connective tissue and collagen will be determined as percent of positive intralobular stain to total lobular area per case. Intralobular connective tissue content will be examined using Hematoxylin and Eosin (H&E) stain and fibrillar collagen content via Masson's trichrome stain.

Isolation and differentiation of human monocyte-derived Mphs: Human Mphs will be differentiated from blood monocytes isolated from the same patient than the tumor sample. Blood samples will be obtained following standard ethical procedures and with the approval of the concerned Internal Review Boards.

Human blood-derived Mphs will be stained with CellTracker™ Green 5-chloromethylfluorescein diacetate (CMFDA) Dye prior to co-culture with breast tumors explants to allow distinguishing them from endogenous Mphs in immunohistochemistry staining.

Ex vivo tumor slice preparation and co-culture with Mphs: Ex vivo tumor slices will be performed. Surgical samples will be embedded in 3% low gelling temperature agarose prepared in Phosphate Buffered Saline (PBS) to allow for easier slicing. 500-µm slices will be obtained with a microtome dedicated to live tissues, a Krumdieck tissue slicer filled with ice-cold PBS set to medium blade and arm speeds. Slices will be cultured on 30-mm cell culture insert featuring a hydrophilic PolyTetraFluoroEthene (PTFE) membrane with pore size of 0.4 µm (Merck Millipore) placed inside 6-well plates containing 1.1 mL of Dulbecco's Modified Eagle Medium (DMEM) with or without Ameboid Migration (AM) or Mensenchymal Migration (MM) inhibitors. The same day, co-cultures will be performed by seeding 5 × 105 human Monocyte Derived Macrophages (hMDMs) on top of tumor slices and left in a 37°C 5% CO2 environment. Culture medium will be replaced daily for three days before overnight fixation with formalin at 4°C (Sigma-Aldrich).

For determination of the Mph migration mode, two parameters will be evaluated to determine the migration mode of Mphs inside tumors: the sensitivity to inhibitors and the cell morphology.Mph will be layered on tumor slices from breast tumor biopsies in the presence or absence of the AM inhibitor (20 µM Y27632) or the MM inhibitor (10 µM Batimastat) to identify the Mph migration mode.

Inhibitors: If the infiltration of Mphs into tissues is inhibited by Y27632 (a ROCK inhibitor) and insensitive to protease inhibitors, and then allow to conclude that they use the AM. If the opposite is true, it will conclude that they use the MM. If inhibitors have an additional effect, it will conclude that both AM and MM are used.

Cell morphology: [Mph have an elongated and protrusive morphology during MM. In contrast, during AM, Mph show a round morphology. Although difficult to assess on ImmunoHistoChemistry (IHC) slices, Mph morphology will be analyzed. If elongated Mph can be detected, it will provide us with additional information to conclude on the migration mode.

Immunohistochemistry on tumor slices: Tumor slices used in co-cultures with hMDMs will be embedded in paraffin. For Mph infiltration quantification assays, slices will then be cut along the diameter and serial sectioning will be performed along the cut. Sections will be stained using an anti-CellTracker™ Green CMFDA Dye Rabbit Polyclonal Antibody (Life technologies) to specifically stain exogeneously added human MDMs. To determine viability of tissue slices, sections will be stained with hematoxylin and eosin to assess cell apoptosis and necrosis. Slides will then be scanned using a Panoramic 250 Flash II slide scanner (3DHISTECH, Hungary) with a 20× magnification lens..The number of Mphs per mm2 of tissues will be quantified (Mirax Scan Zeiss virtual slide scanner). This task will be accomplished withDrTalal Al Saati, supervisor of the experimental histopathology technical platform (INSERM-IFR150/Génopole Toulouse-Midi Pyrénées, CHU Purpan, Toulouse).

Value-creation of experimental results: The Mph migration mode will be identified in a significant number of human primitive breast carcinoma of each type as defined by clinicians, based on their histological type, grade, tumor size, hormone receptor status, HER2 status and index of proliferation and clinical characteristics of the patients collected by team2. Moreover, the migration mode of Mph in the healthy tissue from the same patients will be analysed in parallel and will be used as a reference of Mph migration in non-tumoral tissue in each patients. Then, it will determine i) if Mph perform MM in all types of tumor or if they use MM in some tumors and AM in others, and ii) whether a correlation exists between the migration mode used by macrophages to infiltrate tumors and the type of tumor. Finally, it will establish if there is a correlation between the invasive properties of the studied breast cancer (which will be determined by histo-pathological analysis performed by team2) and the migration mode used by Mph in order to determine whether a correlation exists between the migration mode used by macrophages and tumor invasiveness. Actually, the result expected is that when TAMs use the MM which involves proteases and deep remodeling of the extracellular matrices, the tumor invasiveness will be higher than in tumors in which Tyro-3, Axl, and Mer (TAMs) use the AM.

In the long term, the patient outcome will also be taken into account in these analyses as an additional knowledge about the relationship between TAM migration and tumor progression.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient with breast cancer
2. Age > 18 years old
3. Available primary breast tumor sample with adjacent normal epithelial structures
4. Informed consent obtained and signed

Exclusion Criteria:

1. Primary tumor size < 1cm
2. Surgical tumor sample without available adjacent normal epithelial structures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Analysis of Breast Tumor sample | up to 2 years
  analysis of the sensitivity to inhibitors
Analysis of Breast Tumor sample | up to 2 years
  analysis of the cell morphology

CONTACTS AND LOCATIONS:
Overall Officials: Florence Dalenc, Dr, Principal Investigator — Institut Claudius Regaud

IPD SHARING:
Plan to Share IPD: Yes
Specific data base